CLINICAL TRIAL: NCT04454645
Title: Intervening With Opioid-Dependent Mothers Living in Poverty: Effects on Mothers' and Infants' Behavioral and Biological Regulation
Brief Title: Intervening With Opioid-Dependent MothersMothers and Infants
Acronym: mABC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Mary Dozier, Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: mABC; 1R01HD098525-01A1 (NIH)
Record Dates: First submitted 2020-04-09; First posted 2020-07-01 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Opioid Dependence; Parenting; Infant Development
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified ABC (Experimental): 12-session home visiting intervention designed to increase parental sensitivity and nurturance and decrease parental frightening behavior.
  Interventions: Behavioral: mABC
- Modified DEF (Active Comparator): 12-session home visiting intervention designed to increase parental playful interactions that stimulate infant cognitive and motor development
  Interventions: Behavioral: mDEF

INTERVENTIONS:
Behavioral: mABC — Intervention targets parenting sensitivity and nurturance.
  Arms: Modified ABC
Behavioral: mDEF — Intervention targets parenting enhancing infant cognitive development
  Arms: Modified DEF

SUMMARY:
This study will assess the efficacy of the modified Attachment and Biobehavioral Catch-Up (mABC) Intervention, adapted for use with peripartum mothers receiving medication-assisted treatment for opioid use disorder. The investigators expect that mothers who receive the modified Attachment and Biobehavioral Catch-up Intervention will show more nurturing and sensitive parenting and more adaptive physiological regulation than parents who receive a control intervention. The investigators expect that infants whose mothers receive the modified Attachment and Biobehavioral Catch-up will show better outcomes in attachment, behavior, and physiological regulation than infants of parents who receive the control intervention.

DETAILED DESCRIPTION:
Pregnant mothers will be randomly assigned to receive the modified ABC intervention or the control intervention (modified DEF). Hypotheses relate to parent and child outcomes associated with the intervention. Hypothesis 1: Compared to mothers who receive the control intervention, mothers who receive the mABC intervention will show more nurturing and sensitive parenting, enhanced neural activity during parenting-relevant tasks, and more normative patterns of DNA methylation, autonomic nervous system activity, and cortisol production. Hypothesis 2: Compared to infants of mothers who receive the control intervention, infants of mothers who receive the mABC intervention will show more organized and secure attachment patterns, better behavioral regulation during stressors, more advanced social-emotional development, and more normative patterns of DNA methylation, autonomic nervous system activity, and cortisol production. Hypothesis 3: Enhanced maternal sensitivity will mediate effects of the mABC intervention on improved infant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Opioid-dependent pregnant women in third trimester of pregnancy on medication-assisted treatment

Exclusion Criteria:

* None

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Maternal sensitivity | Pre-intervention (3rd trimester)
  The mother will be assessed interacting with the infant simulator. Parental sensitivity (a composite of following the child's lead in interactions, providing nurturance when the child is distressed, and showing positive regard) will be assessed using procedures and coding from the assessment used by the NICHD Study of Early Child Care and Youth Development (Brady-Smith et al., 1999). Sensitivity will be assessed on a 5-point scale with higher scores indicating greater sensitivity.
Maternal sensitivity | Infant age of 3 months
  The mother will be assessed interacting one-to-one with her infant. Parental sensitivity (a composite of following the child's lead in interactions, providing nurturance when the child is distressed, and showing positive regard) will be assessed using procedures and coding from the assessment used by the NICHD Study of Early Child Care and Youth Development (Brady-Smith et al., 1999). Sensitivity will be assessed on a 5-point scale with higher scores indicating greater sensitivity.
Maternal sensitivity | Infant age of 6 months
  The mother will be assessed interacting one-to-one with her infant. Parental sensitivity (a composite of following the child's lead in interactions, providing nurturance when the child is distressed, and showing positive regard) will be assessed using procedures and coding from the assessment used by the NICHD Study of Early Child Care and Youth Development (Brady-Smith et al., 1999). Sensitivity will be assessed on a 5-point scale with higher scores indicating greater sensitivity.
Maternal sensitivity | Infant age of 12 months
  The mother will be assessed interacting one-to-one with her infant. Parental sensitivity (a composite of following the child's lead in interactions, providing nurturance when the child is distressed, and showing positive regard) will be assessed using procedures and coding from the assessment used by the NICHD Study of Early Child Care and Youth Development (Brady-Smith et al., 1999). Sensitivity will be assessed on a 5-point scale with higher scores indicating greater sensitivity.
Maternal methylation of μ-opioid receptor (OPRM1) gene | Pre-intervention (3rd trimester)
  Maternal methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva
Maternal methylation of μ-opioid receptor (OPRM1) gene | Infant age of 12 months
  Maternal methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva
Maternal methylation of oxytocin receptor (OXTR) gene | Pre-intervention (3rd trimester)
  Maternal methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva
Maternal methylation of oxytocin receptor (OXTR) gene | Infant age of 12 months
  Maternal methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva
Infant methylation of μ-opioid receptor (OPRM1) gene | Pre-intervention (3rd trimester)
  Infant methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva
Infant methylation of μ-opioid receptor (OPRM1) gene | Infant age of 12 months
  Infant methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva
Maternal neural activity (Event related potentials - ERP) - Own child-other child task | Pre-intervention (3rd trimester)
  Maternal event-related potentials (ERP) will be assessed while viewing photos of their own infants, familiar infants, and unfamiliar infants. The P300 (a positive deflection about 300 ms after the stimuli) will be studied, with a bigger difference between own and other child considered preferable.
Maternal neural activity (Event related potentials - ERP) - Own child-other child task | Infant age of 12 months
  Maternal event-related potentials will be assessed while viewing photos of their own infants, familiar infants, and unfamiliar infants. The P300 (a positive deflection about 300 ms after the stimuli) will be studied, with a bigger difference between own and other child considered preferable.
Maternal neural activity (Event related potentials - ERP) - Reward sensitivity task | Pre-intervention (3rd trimester)
  Maternal event-related potentials will be assessed while viewing images from four categories: opioid-related images, baby pictures, positive images, and neutral images. The P300 (a positive deflection about 300 ms after the stimuli) will be studied, with a bigger difference between child and opioid-related images considered preferable.
Maternal neural activity (Event related potentials - ERP) - Reward sensitivity task | Infant age of 12 months
  Maternal event-related potentials will be assessed while viewing images from four categories: opioid-related images, baby pictures, positive images, and neutral images. The P300 (a positive deflection about 300 ms after the stimuli) will be studied, with a bigger difference between child and opioid-related images considered preferable.
Maternal neural activity (Event related potentials - ERP) - Child emotion task | Pre-intervention (3rd trimester)
  Maternal event-related potentials will be assessed while viewing images of children crying, laughing, and showing neutral expressions. The N180 (a negative deflection about 180 ms after the stimuli) will be studied, with a bigger difference between faces will be considered preferable.
Maternal neural activity (Event related potentials - ERP) - Child emotion task | Infant age of 12 months
  Maternal event-related potentials will be assessed while viewing images of children crying, laughing, and showing neutral expressions. The N180 (a negative deflection about 180 ms after the stimuli) will be studied, with a bigger difference between faces will be considered preferable.
Maternal parasympathetic nervous system activity during Still Face | Pre-intervention (3rd trimester)
  The control of cardiac functions via the vagal nerve, or vagal tone, is an index of parasympathetic activity. It can be measured by heart rate variability associated with respiration or high frequency respiratory sinus arrhythmia (RSA). RSA data will be collected continuously throughout a 15-minute period during the Still Face Procedure using a MindWare Portable Lab system. Greater changes in RSA from baseline to still face considered preferable.
Maternal parasympathetic nervous system activity | Infant age of 12 months
  The control of cardiac functions via the vagal nerve, or vagal tone, is an index of parasympathetic activity. It can be measured by heart rate variability associated with respiration or high frequency respiratory sinus arrhythmia (RSA). RSA data will be collected continuously throughout a 15-minute period during the Still Face Procedure using a MindWare Portable Lab system. Greater changes in RSA from baseline to still face considered preferable.
Infant parasympathetic nervous system activity | Infant age of 6 months
  The control of cardiac functions via the vagal nerve, or vagal tone, is an index of parasympathetic activity. It can be measured by heart rate variability associated with respiration or high frequency respiratory sinus arrhythmia (RSA). RSA data will be collected continuously throughout a 15-minute period during the Still Face Procedure using a MindWare Portable Lab system. Greater changes in RSA from baseline to still face considered preferable.
Infant parasympathetic nervous system activity | Infant age of 12 months
  The control of cardiac functions via the vagal nerve, or vagal tone, is an index of parasympathetic activity. It can be measured by heart rate variability associated with respiration or high frequency respiratory sinus arrhythmia (RSA). RSA data will be collected continuously throughout a 15-minute period during the Still Face Procedure using a MindWare Portable Lab system. Greater changes in RSA from baseline to still face considered preferable.
Infant diurnal cortisol production | Infant age of 6 months
  Infant diurnal cortisol production will be assessed through salivary cortisol levels collected at waketime and bed-time.
Infant diurnal cortisol production | Infant age of 12 months
  Infant diurnal cortisol production will be assessed through salivary cortisol levels collected at waketime and bed-time.
Infant behavioral regulation | Infant age of 6 months
  Behavioral coding of emotion regulation will be conducted from video recordings of the Still Face Paradigm on the Behavioral Regulation Scale, a mild social stressor. Behavior regulation will be coded on a scale called Behavior Regulation. The scores will be continuous with higher scores indicating better regulation (ranging from 1-9).
Infant behavioral regulation | Infant age of 12 months
  Behavioral coding of emotion regulation will be conducted from video recordings of the Still Face Paradigm on the Behavioral Regulation Scale, a mild social stressor. Behavior regulation will be coded on a scale called Behavior Regulation. The scores will be continuous with higher scores indicating better regulation (ranging from 1-9).
Infant attachment | Infant age of 12 months
  Infant attachment will be assessed using the Strange Situation. Coding will be completed using the standard Strange Situation coding scheme (with 4 major categories, with secure preferable).
Infant cognitive development | Infant age of 12 months
  Infant cognitive development will be assessed through maternal report on the Ages and Stages Questionnaire. Scores could range from 0-300 with higher scores reflecting higher functioning.

SECONDARY OUTCOMES:
Maternal substance use | Pre-intervention (3rd trimester)
  Mothers will report on substance use through the Timeline Follow-Back Interview. Higher scores will reflect more use of illicit substances (score from 0-unlimited).
Maternal substance use | Infant age of 12 months
  Mothers will report on substance use through the Timeline Follow-Back Interview. Higher scores will reflect more use of illicit substances (score from 0-unlimited).
Maternal depression | Pre-intervention (3rd trimester)
  Mothers will report on their depression on the Beck Depression Inventory - II, with higher scores indicating more depressive symptoms reported. (Scores could range from 0-63.)
Maternal depression | Infant age of 12 months
  Mothers will report on their depression on the Beck Depression Inventory - II, with higher scores indicating more depressive symptoms reported. (Scores could range from 0-63.)
Maternal executive functioning | Pre-intervention (3rd trimester)
  Mothers will complete Flanker task. Scores have a mean of 100 with a standard deviation of 15, with higher scores reflecting stronger executive functioning.
Maternal executive functioning | Infant age of 12 months
  Mothers will complete Flanker task. Scores have a mean of 100 with a standard deviation of 15, with higher scores reflecting stronger executive functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Dozier, Ph.D., Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States